CLINICAL TRIAL: NCT07134673
Title: Mitochondrial Oxygen Consumption and Substrate Utilisation In Vitro in Peripheral Blood Mononuclear Cells, and In Vivo on Muscle and Skin in Long COVID Patients and Convalescent Individuals: A Case-Control and Diagnostic Accuracy Study
Brief Title: Mitochondrial Function in Peripheral Blood Mononuclear Cells, Muscle, and Skin of Long COVID Patients
Acronym: MitoLoCo
Status: Not yet recruiting | Type: Observational
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Principal Investigator, Elisabeth De Waele, Head of the Department of Clinical Nutrition, Co-director of Vitality Research Group, Universitair Ziekenhuis Brussel
Other Study IDs: EC-2025-071; G075423N (Other: Vrije Universiteit Brussel, Universitair Ziekenhuis Brussel)
Record Dates: First submitted 2025-06-25; First posted 2025-08-21 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Long COVID; Post-COVID-19 Condition
Keywords: mitochondrial dysfunction
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; Mitochondrial Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral Blood Mononuclear Cells
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Individuals with long COVID: History of a confirmed or documented SARS-CoV-2 infection and long COVID according to the World Health Organisation's clinical case definition
- Convalescent individuals: History of a confirmed or documented SARS-CoV-2 infection, complete recovery after the SARS-CoV-2 infection, no history of long COVID according to the World Health Organisation's clinical case definition

SUMMARY:
Mitochondria are structures inside cells that are responsible for producing energy from nutrients through a series of steps, using oxygen. To have an idea of how well the mitochondria can produce energy, we can measure how much oxygen they use. The goal of this study is to:

1. To compare the oxygen use between people with long COVID and people who completely recovered after COVID-19, using three techniques that measure the oxygen use in blood cells, on the skin and in the muscle
2. To test how similar these three techniques are in measuring the oxygen used in the three different tissues

Participants will:

* Complete surveys,
* Wear an activity tracker (7 days),
* Undergo several non-invasive tests, and
* Donate a blood sample The study will take place in UZ Brussel hospital and will take 2 study visits, approximately 7 days apart.

ELIGIBILITY:
Individuals with long COVID:

Inclusion criteria:

* Long COVID diagnosis, based on the WHO definition;
* Presence of long COVID symptoms for a minimum of 6 months.
* History of confirmed or documented SARS-CoV-2 infection.
* Adult (≥18 years of age).
* Post-COVID-19 Functional Status Scale grade 2-4, while they had a grade 0 before the SARS-CoV-2 infection.

Exclusion criteria:

* Pre-existing chronic diseases potentially affecting the functional status scale.
* Treatment with metabolism altering drugs.
* > 10 standard units of alcohol (10 grams of alcohol/glass) per week.
* Unable to understand oral and written instructions in Dutch, French or English.
* Allergies to medical adhesive bandages.
* Porphyria and other skin conditions aggravated by sunlight.

Convalescent individuals

Inclusion criteria:

* History of confirmed or documented SARS-CoV-2 infection.
* Complete recovery after the SARS-CoV-2 infection, no history of long COVID based on the WHO definition;
* Post-COVID-19 Functional Status Scale [2] grade 0 both before the infection and currently.
* Adult (≥18 years of age).

Exclusion criteria:

* Pre-existing chronic non-communicable diseases (e.g. hypertension, chronic respiratory diseases, diabetes).
* Treatment with metabolism altering drugs.
* > 10 standard units of alcohol (10 grams of alcohol/glass) per week.
* Unable to understand oral and written instructions in Dutch, French or English.
* Allergies to medical adhesive bandages.
* Porphyria and other skin conditions aggravated by sunlight.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study participants will be recruited in the Universitair Ziekenhuis Brussel, from the general population in Belgium through traditional and social media, as well as in the vicinity of the study site through leaflets and posters.
Sampling Method: Non-Probability Sample
Enrollment: 54 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Basal Oxygen Consumption rate (pmol O2/min) | Blood sample is taken during the second study visit (approximately 7 days after the first study visit) and the PBMCs are cryopreserved until analysis (after all participants have been recruited, estimated to be within 1 year of the start of the study)
  Seahorse XF Substrate Oxidation Stress test analysis of the peripheral blood mononuclear cells (PBMCs)
Tissue Saturation Index (TSI) | Second study visit (approximately 7 days after the first study visit)
  Near-infrared spectroscopy
Mitochondrial oxygen tension (mitoPO2) (mmHg/s) | Second study visit (approximately 7 days after the first study visit)
  Cellular Oxygen Metabolism monitoring
Mitochondrial oxygen consumption (mitoVO2) | Second study visit (minimally 7 days after the first study visit)
  Cellular Oxygen Metabolism monitoring

SECONDARY OUTCOMES:
Proportion of participants meeting the criteria for PEM | Second study visit (minimally 7 days after the first study visit)
  De Paul Symptom Questionnaire - Post-exertional malaise (DSQ-PEM)
General fatigue | Second study visit (approximately 7 days after the first study visit)
  Multidimensional Fatigue Inventory (MFI-20)
Physical fatigue | Second study visit (approximately 7 days after the first study visit)
  Multidimensional Fatigue Inventory (MFI-20)
Mental fatigue | Second study visit (approximately 7 days after the first study visit)
  Multidimensional Fatigue Inventory (MFI-20)
Reduced activities | Second study visit (approximately 7 days after the first study visit)
  Multidimensional Fatigue Inventory (MFI-20)
Reduced motivation | Second study visit (approximately 7 days after the first study visit)
  Multidimensional Fatigue Inventory (MFI-20)
Severity and impact of fatigue on daily life | Second study visit (approximately 7 days after the first study visit)
  The Fatigue Severity Scale (FSS) contains nine statements that rate the severity of the fatigue symptoms. The statements are rated from 1 to 7, with a low value indicating strong disagreement with the statement and a high value indicating strong agreement with the statement. The total score is the sum of the individual scores, with a higher score indicating a greater impact of fatigue on daily life.
Symptom burden (θ) | First study visit
  Item Response Theory (IRT) will be applied to estimate a latent trait representing symptom burden, using Section 2.6 of the WHO Post-COVID-19 Case Report Form. Symptoms will be coded as binary variables (1 = symptom present, 0 = symptom absent). IRT modeling will be used to derive a latent trait estimate (θ) for each individual, reflecting the overall severity or burden of symptoms.
Resting Energy Expenditure (kcal/kg body weight/day) | Second study visit (approximately 7 days after the first study visit)
  Indirect calorimetry will be used to measure the Resting Energy Expenditure (kcal/day). This value will be divided by the body weight (kg) on that same day.
Basal Oxygen Consumption rate (pmol O2/min) | Blood sample is taken during the second study visit (approximately 7 days after the first study visit) and the PBMCs are cryopreserved until analysis (after all participants have been recruited, estimated to be within 1 year of the start of the study)
  Seahorse XF Substrate Oxidation Stress test analysis of the peripheral blood mononuclear cells (PBMCs) after substrate pathway inhibitor Etomoxir is used
Basal Oxygen Consumption rate (pmol O2/min) | Blood sample is taken during the second study visit (approximately 7 days after the first study visit) and the PBMCs are cryopreserved until analysis (after all participants have been recruited, estimated to be within 1 year of the start of the study)
  Seahorse XF Substrate Oxidation Stress test analysis of the peripheral blood mononuclear cells (PBMCs) after substrate pathway inhibitor UK5099 is used
Basal Oxygen Consumption rate (pmol O2/min) | Blood sample is taken during the second study visit (approximately 7 days after the first study visit) and the PBMCs are cryopreserved until analysis (after all participants have been recruited, estimated to be within 1 year of the start of the study)
  Seahorse XF Substrate Oxidation Stress test analysis of the peripheral blood mononuclear cells (PBMCs) after substrate pathway inhibitor BPTES is used
Maximal Oxygen Consumption rate (pmol O2/min) | Blood sample is taken during the second study visit (approximately 7 days after the first study visit) and the PBMCs are cryopreserved until analysis (after all participants have been recruited, estimated to be within 1 year of the start of the study)
  Seahorse XF Substrate Oxidation Stress Test analysis of the peripheral blood mononuclear cells (PBMCs) after substrate pathway inhibitor Etomoxir is used
Maximal Oxygen Consumption rate (pmol O2/min) | Blood sample is taken during the second study visit (approximately 7 days after the first study visit) and the PBMCs are cryopreserved until analysis (after all participants have been recruited, estimated to be within 1 year of the start of the study)
  Seahorse XF Substrate Oxidation Stress Test analysis of the peripheral blood mononuclear cells (PBMCs) after substrate pathway inhibitor UK5099 is used
Maximal Oxygen Consumption rate (pmol O2/min) | Blood sample is taken during the second study visit (approximately 7 days after the first study visit) and the PBMCs are cryopreserved until analysis (after all participants have been recruited, estimated to be within 1 year of the start of the study)
  Seahorse XF Substrate Oxidation Stress Test analysis of the peripheral blood mononuclear cells (PBMCs) after substrate pathway inhibitor BPTES is used
Respiratory Quotient | Second study visit (approximately 7 days after the first study visit)
  Indirect calorimetry

OTHER OUTCOMES:
Weight (kg) | Second study visit (approximately 7 days after the first study visit)
  Body weight (kg) in light indoor clothes without shoes.

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth De Waele, MD. PhD., Principal Investigator — Vitality Research Group, Metabolism and Nutrition, Vrije Universiteit Brussel (VUB), Clinical Nutrition Department, Universitair Ziekenhuis Brussel (UZ Brussel)
Locations (1):
- Laarbeeklaan 101, Jette, Brussels Capital, Belgium

IPD SHARING:
Plan to Share IPD: Undecided
Based on the guidelines and regulations of the Vrije Universiteit Brussel, the IPD will be shared. Plan is yet to be determined.